CLINICAL TRIAL: NCT04819750
Title: Impact of Music Therapy on Intraoperative Patient Comfort During Cataract Surgery With Topic Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MUSICOTOPICAT
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Cataract; Anxiety
MeSH Terms: conditions — Cataract; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MusicCare® device (Active Comparator): The device is a touch tablet with a headset that allows noise reduction. The patient can choose the music they prefer. The selected U-shaped sequence uses the principles of hypnoanalgesia to accompany the patient into a state of deep relaxation.
  Interventions: Device: MusicCare® device
- Headphones with noise reduction (Placebo Comparator): Headphones with noise reduction without music
  Interventions: Device: Headphones with noise reduction

INTERVENTIONS:
Device: MusicCare® device — The device is a touch tablet with a headset that allows noise reduction. The patient can choose the music they prefer. The selected U-shaped sequence uses the principles of hypnoanalgesia to accompany the patient into a state of deep relaxation.
  Arms: MusicCare® device
Device: Headphones with noise reduction — Headphones with noise reduction without music
  Arms: Headphones with noise reduction

SUMMARY:
Cataract surgery with topic anesthesia is anxiety provoking. This operative stress can increase pain perception and blood pressure. This discomfort can lead to non-compliance with immobility and potentially lead to intraoperative and postoperative complications.

Pharmacological means are limited to reduce anxiety. Only anxiolytics could be effective but at the cost of side effects not compatible with surgery.

Music Care is a "digital treatment" allowing the diffusion of music with a U-shaped sequence using the principles of hypnoanalgesia.

The objective of this study is to evaluate the effectiveness of the MusicCare listening device on the anxiety of patients during cataract surgery with topic anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Cataract surgery with topical anesthesia

Exclusion Criteria:

* Hearing impaired patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Self-assessed anxiety score between the 2 groups | Baseline day, when entering the operating room
  Self-assessed anxiety score on a visual analogue scale (VAS) from 0 to 10 (0 means no anxiety and 10 the maximum anxiety)

SECONDARY OUTCOMES:
Self-assessment of the duration of the surgery | Baseline day, when entering the operating room
  Self-rated duration of surgery on a scale of 0 to 5 (0 means 5 to 10 minutes and 5 means 25 to 30 minutes)